CLINICAL TRIAL: NCT05888155
Title: Clinical Presentation of Genetic Disorders in Patients Attending Genetic Outpatient Clinic of Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Ali Soliman Mohammed, Doctor, Assiut University
Other Study IDs: Genetic disorders presentation
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Genetic Disease Clinical Presentation in Patients Attending Genetics Outpatient Clinic of Assiut University Children Hospital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genetic Epidemiology : is quickly expanding research field concerned with considerate the heritable aspect of disease risk, individual propensity to disease and eventually with contributing to a complete molecular understanding of pathogenesis. Genetics : is the scientific study of genes &heredity of how certain qualities or traits are passed from parents to offspring as a result of changes in DNA sequence . A gene is a segment of DNA that contains instructions for building of one or more molecules Genetic disorders: is a health problem caused by one or more abnormalities in the genome. It can be caused by a mutation in a single gene (monogenic) or multiple genes (polygenic) or by a chromosomal abnormality. (1)mutations: affect the human genes either inherited from one or both parents or due to certain environmental factors Four of the main types include:(1)Single _gene inheritance diseases :Single gene inheritance diseases are diseases that occur because one defective gene is present. They are known as monogenetic disorders.(EX:Marfan Syndrome ) (2)Multifactorial genetic inheritance disorders : Genetic disorders may also be complex, , meaning they are likely associated with the effects of multiple genes in combination with lifestyles and environmental factors. Multifactorial disorders include heart disease and diabetes. (3)chromosomal abnormalities : result from a problem with cell division and arise because of duplications or absences of entire chromosomes or pieces of chromosomes. Examples of chromosome abnormality disorders include(Down sydrome ) (4)Mitochondrial genetic inheritance disorders : are caused by mutations in the DNA of mitochondria, small particles within cell. Mitochondrial DNA is always inherited from the female parent since egg cells (unlike sperm cells) keep their mitochondrial DNA during the process of fertilization. Environmental Factors: called (mutagens)which can lead to genetic mutations Such as Chemical exposure , Radiation exposure , Smoking , UV rays exposure from the sun prognosis Of genetic disorders: Not all genetic disorders directly result in death, there are no known cures for genetic disorders. Many genetic disorders affect stages of development, such as Down syndrome, while others result in purely physical symptoms such as muscular dystrophy. Other disorders, such as Huntington's disease, show no signs until adulthood. .Treatment of genetic disorders: The treatment of genetic disorders is an ongoing battle, with over 1,800 gene therapy clinical trials having been completed, are ongoing, or have been approved worldwide, Despite this, most treatment options revolve around treating the symptoms of the disorders in an attempt to improve patient quality of life. Diagnosis of genetic disorders: (1)personal medical history :information about an individual health often going back to birth can provide clues to a genetic diagnosis (2)physical examination :certain physical characteristics , such as distinctive facial features can suggest the diagnosis of a genetic disorder , a geneticist will do a through physical Examination that may include measurements such as head circumference and so on . (3) Family health history :because genetic conditions often run in families , information about the health of family members can be a critical tool for diagnosing these disorders . (4)Laboratory Tests :including genetic testing , molecular , chromosomal , and biochemical genetic or genomic testing are used to diagnose genetic disorders. Genetic counselling is a communication process, which aims to help individuals, couples and families understand and adapt to the medical, psychological, familial and reproductive implications of the genetic contribution to specific health conditions. Patients With History Of TORCH: Bad Obstetric history (BOH) implies previous unfavorable foetal outcome in terms of two or more consecutive spontaneous abortion, history of intrauterine foetal death, intrauterine growth retardation, still births, early neonatal death and/or congenital anomalies. Cause of BOH may be genetic, hormonal, abnormal maternal immune response and maternal infection.

DETAILED DESCRIPTION:
A descriptive study to determine the clinical presentation of patients attending Assiut University children hospital and availability of investigations can be done for them .

ELIGIBILITY:
Inclusion Criteria:

- The study will include all infants &children(from age of one day to age of 18 years ) attending Assiut University children hospital with symptoms suggesting genetic disorders

Exclusion Criteria:

* No

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All infants & children from age of one day to age of 18 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Clinical presentation of genetic disorders in patients attending genetics outpatient clinic of Assiut university children hospital | One year
  Detection of clinical presentation of genetic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Ahmed Mahmoud, Doctor, Study Director — Assiut University; Zeinab Mohamed Mohi_eldin, Doctor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] MidlinePlus.gov:Medlineplus(internet) .Bethesda (MD)National library of medicine (US)(updated june24)cited (2020Jul 1.)
- [Background] Cavazzano human beta-- Calvo, M. (2010). Transfusion thalassaemia. Nature 467, 318independence and HMGA2 activation after gene therapy of 322. doi:10.1038/nature09328 Cideciyan, A.V. et al (22 January 2013). Human retinal gene therapy for Leber congenital amaurosis shows advancing retinal de generation despite enduring visual improvement. Proceedings of the National Academy of Sciences of the United States of America, Earline Online Publication. doi: 10.1073/pnas.1218933110 MacLaren, R.E. et al (16 January 2014). Retinal gene therapy in patien ts with choroideremia: initial findings from a phase 1/2 clinical trial. The Lancet, Early Online Publication. doi:10.1016/S01406736(13)62117 Nathwani, A.C. (2011). Adenovirusassociated virus vector-- 0 mediated gene transfer in hemophilia B. The New Engla nd Journal of Medicine, 365(25), 23572365. Nienhuis, A.W. (2013). Development of gene therapy for blood disorders: an update. Blood 122(9), 1556 1564. doi: 10.1182/blood201304453209 Palfi, S. et al (10 January 2014). Longterm safety and tolerability o f ProSavin, a lentiviral vector-- based gene therapy for parkinson's disease; a dose escalation, open Publication. doi: 10.1016/S014006736(13)61939Xlabel, phase 1/2 trial. The Lancet, Early Online Penn Medicine (7 December 2013). Penn medicine team reports findings from research study of first 59 adult and pediatric leukemia patients who received investigational, personalized cellular therapy CTL019. Retrieved from http://www.uphs.upenn.edu/news/News_Releases/2013/12/ctl019/ Persons, Derek A. (2010). Gene t 10.1038/467277a Petrsherapy: Targeting betathalassaemia. Nature 467, 277278. doi: Silva, H. & R. Linden (2014). Advances in gene therapy technologies to treat retinitis pigmentosa.
- [Background] 3)National Human genome Research Institute; Led by Director Eric Green, M.D., Ph.D., the National Human Genome Research Institute (NHGRI) is the driving force for advancing genomics research at the National Institutes of Health (NIH), the largest biomedical research agency in the world. (18/5/2018)
- [Background] Garvan Institute of Medical Research/an Australian biomedical research institute located in Darlinghurst, Sydney, New South Wales/ directed by professor Chris Goodnow , FAA, FRS.
- [Result] National Institute of General Medical Sciences (301_496_7301): Supports basic research that increase understanding of biological processes&lays the foundation for advances in disease diagnosis, treatment&prevention.
- Available data/document: Clinical Study Report: 01095697530 — http://Shaimaa4796@gmail.com